CLINICAL TRIAL: NCT07382908
Title: A Single-Center, Single-Dose, Randomized, Open-Label, Single-Period, Parallel Bioequivalence Study of BGM0504 Injection in Overweight/Obese Participants
Brief Title: Bioequivalence Study of BGM0504 Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Collaborators: BrightGene Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGM0504-BE
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Overweight/Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — penclomedine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: BGM0504 Injection multi-dose pen
- Group B (Experimental)
  Interventions: Drug: BGM0504 Injection single-dose pen
- Group C (Active Comparator)
  Interventions: Drug: BGM0504 Injection single-dose pen

INTERVENTIONS:
Drug: BGM0504 Injection multi-dose pen — 5 mg, single subcutaneous injection in the abdominal region
  Arms: Group A
Drug: BGM0504 Injection single-dose pen — 5 mg, single subcutaneous injection in the abdominal region
  Arms: Group B
Drug: BGM0504 Injection single-dose pen — 5 mg, single subcutaneous injection in the abdominal region
  Arms: Group C

SUMMARY:
This is a study to evaluate the bioequivalence of a single subcutaneous injection of BGM0504 multi-dose pen (experimental formula T1) and BGM0504 single-dose pen (experimental formula T2) with BGM0504 single-dose pen (reference formula R).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years (inclusive).
* Male weight ≥50 kg, female weight ≥45 kg, and overweight (24.0 ≤ BMI < 28.0 kg/m²) or obese (BMI ≥ 28.0 kg/m²).
* From signing the ICF until 3 months after dosing, no pregnancy plan and willing to use effective contraception to avoid pregnancy or causing partner pregnancy, and no plan for sperm/egg donation.
* The participant fully understands the trial purpose, nature, methods, and potential adverse reactions, can complete the trial according to the protocol, has good living habits, can maintain good communication with the investigator, and voluntarily signs the ICF.

Exclusion Criteria:

* History of severe allergies or severe specific allergic diseases/history (asthma, urticaria, eczematous dermatitis, etc.) or allergic constitution (allergic to two or more foods or drugs), known or suspected allergy to any excipient of BGM0504 Injection.
* Previous diagnosis of type 1 or type 2 diabetes, or clinically significant abnormal HbA1c at screening.
* Family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 syndrome.
* History of acute/chronic pancreatitis, pancreatic injury, or other high-risk factors for pancreatitis.
* Past or screening findings of digestive system diseases that may increase participant risk.
* Positive for HBsAg, HCV antibody, syphilis antibody, or HIV antibody at screening.
* Participation in any drug or medical device clinical trial and receiving investigational product/device intervention within 3 months prior to screening.
* Consumption or plan to consume specific foods (including pitaya, mango, grapefruit, pomelo or their juices, high-purine foods like animal organs, seafood, chocolate) or beverages containing caffeine/alcohol within 48 hours before dosing; or unwilling to stop consuming these during the in-house period.
* Pregnant or breastfeeding women, or positive pregnancy test at screening.
* Any other condition considered by the investigator as unsuitable for participation or participant withdrawal due to personal reasons..

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0 to 672 hours
  Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 0 to 672 hours
  Area under the plasma concentration versus time curve (AUC)0-t

SECONDARY OUTCOMES:
Monitor all the adverse event | 29 days
  Monitor all the adverse event was assessed by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China